CLINICAL TRIAL: NCT02721836
Title: Randomized Controlled Trial on Yoga for Irritable Bowel Syndrome
Brief Title: Yoga for Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Dania Schumann, Principal Investigator, Research fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-6653-BO
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): 12 week yoga course, two times a week 75 minutes each time
  Interventions: Behavioral: Yoga
- Nutrition (Active Comparator): 3 counselling sessions within 12 weeks
  Interventions: Behavioral: Nutrition Counselling

INTERVENTIONS:
Behavioral: Yoga — Yoga intervention 12 weeks, twice weekly 75-minute intervention Yoga postures, breathing, relaxation, and meditation
  Arms: Yoga
Behavioral: Nutrition Counselling — Evidence-based Nutrition Counselling, 3 appointments within 12 weeks
  Arms: Nutrition

SUMMARY:
The proposed study aims to investigate the feasibility, effectiveness, and perceived benefit of a hatha yoga intervention for patients with irritable bowel syndrome (IBS) compared to nutrition counselling. Further, the potential of both interventions to influence the gut microbiome will be inquired.

ELIGIBILITY:
Inclusion Criteria:

* Patients with irritable bowel syndrome (IBS) diagnosed by physician and confirmed by Rome III diagnostic criteria

Exclusion Criteria:

* inflammatory bowel diseases (IBD)
* total abdominal colectomy
* no sonographie or colonoscopy as diagnostic criterion
* stool lactoferrin > 7mg/g
* pregnancy or breast feeding
* simultaneous participation in further clinical intervention trials
* Regular yoga practice or nutrition counselling in the past 12 months
* Planned surgery in the study period
* Serious illness that would interfere with the ability to practice yoga

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptoms | Week 12
  Irritable Bowel Syndrome Severity Scoring System (IBS-SSS)

SECONDARY OUTCOMES:
disease specific quality of life | Week 12
  Irritable Bowel Syndrome Quality of Life measurement (IBS-QOL)
disease specific quality of life | Week 24
  Irritable Bowel Syndrome Quality of Life measurement (IBS-QOL)
Generic Health-related Quality of life | Week 12
  Short Form 36 Health Survey Questionnaire, SF-36
Generic Health-related Quality of life | Week 24
  Short Form 36 Health Survey Questionnaire, SF-36
Emotional distress | Week 12
  Hospital Anxiety and Depression Scale (HADS)
Emotional distress | Week 24
  Hospital Anxiety and Depression Scale (HADS)
Subjective Stress | Week 12
  Cohen Perceived Stress Scale (CPSS)
Subjective Stress | Week 24
  Cohen Perceived Stress Scale (CPSS)
Subjective improvement of symptoms | Week 12
  Adequate Relief Score and Global Improvement Scale (GI)
Subjective improvement of symptoms | Week 24
  Adequate Relief Score and Global Improvement Scale (GI)
Gut microbiome | Week 12
  Stool samples
Adverse Event | Week 12
Adverse Event | Week 24
Irritable Bowel Syndrome Symptoms | Week 24
  Irritable Bowel Syndrome Severity Scoring System (IBS-SSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Universität Duisburg-Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schumann D, Anheyer D, Lauche R, Dobos G, Langhorst J, Cramer H. Effect of Yoga in the Therapy of Irritable Bowel Syndrome: A Systematic Review. Clin Gastroenterol Hepatol. 2016 Dec;14(12):1720-1731. doi: 10.1016/j.cgh.2016.04.026. Epub 2016 Apr 22. PMID 27112106